CLINICAL TRIAL: NCT01871766
Title: Risk-Adapted Focal Proton Beam Radiation and/or Surgery in Patients With Low, Intermediate and High Risk Rhabdomyosarcoma Receiving Standard or Intensified Chemotherapy
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RMS13; NCI-2013-00913 (Registry Identifier: NCI Clinical Trial Registration Program)
Record Dates: First submitted 2013-05-30; First posted 2013-06-07 (Estimated); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Rhabdomyosarcoma
Keywords: Rhabdomyosarcoma; Radiation therapy; Proton beam
MeSH Terms: conditions — Rhabdomyosarcoma | interventions — Vincristine; Dactinomycin; Cyclophosphamide; Surgical Procedures, Operative; Radiation; Proton Therapy; Brachytherapy; Bevacizumab; Vascular Endothelial Growth Factor A; Sorafenib; Granulocyte Colony-Stimulating Factor; Filgrastim; pegfilgrastim; Irinotecan; Ifosfamide; Etoposide; etoposide phosphate; Doxorubicin; Dexrazoxane; Contrast Media

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Low-Risk, Subset 1 (Experimental): Lymph node sampling will take place pretreatment and pre-surgery. Participants receive 12 weeks of chemotherapy (vincristine, dactinomycin and cyclophosphamide). They are then evaluated to determine how the tumor responded to treatment. Twelve additional weeks of chemotherapy (vincristine and dactinomycin) is given, followed by evaluation for tumor response. No further treatment is given, and participants are observed closely. Myeloid growth factor is given if needed.
  Participants also receive ^1^1C-methionine as described in the intervention section.
  Interventions: Drug: Vincristine; Drug: Dactinomycin; Drug: Cyclophosphamide; Procedure: Surgical Resection; Procedure: Radiation; Drug: Myeloid Growth Factor; Procedure: Lymph Node Sampling; Drug: ^1^1C-methionine
- Low-Risk, Subset 2 (Experimental): Lymph node sampling will take place pretreatment and pre-surgery. Participants receive 12 weeks of chemotherapy (vincristine, dactinomycin, cyclophosphamide). The tumor is evaluated to determine how it responded to treatment. Radiation therapy and/or surgical resection is performed to destroy or remove the remaining tumor. Twelve additional weeks of chemotherapy (vincristine, dactinomycin, cyclophosphamide) is given, followed by evaluation for tumor response. If delayed for medical reasons, radiation therapy and/or surgical resection is done at this time. Participants then receive 16 weeks of additional chemotherapy (vincristine, dactinomycin and cyclophosphamide). No further treatment is given, and participants are observed closely. Myeloid growth factor will be given if needed.
  Participants also receive ^1^1C-methionine as described in the intervention section.
  Interventions: Drug: Vincristine; Drug: Dactinomycin; Drug: Cyclophosphamide; Procedure: Radiation; Drug: Myeloid Growth Factor; Procedure: Lymph Node Sampling; Drug: ^1^1C-methionine
- Intermediate-Risk (Experimental): Lymph node sampling takes place pretreatment and pre-surgery. Participants receive 12 weeks of chemotherapy (vincristine, dactinomycin, cyclophosphamide). The tumor is evaluated for treatment response. Radiation therapy and/or surgical resection is done. Twelve weeks of chemotherapy (vincristine, dactinomycin, cyclophosphamide) is followed by evaluation for tumor response. If delayed for medical reasons, radiation therapy and/or surgical resection is done at this time. Participants receive 16 weeks of chemotherapy (vincristine, dactinomycin, cyclophosphamide) followed by 12 weeks of maintenance treatment (bevacizumab, sorafenib, oral cyclophosphamide). No further treatment is given, and participants are observed closely. Myeloid growth factor is given if needed.
  Participants also receive ^1^1C-methionine as described in the intervention section.
  Interventions: Drug: Vincristine; Drug: Dactinomycin; Drug: Cyclophosphamide; Procedure: Surgical Resection; Procedure: Radiation; Drug: Bevacizumab; Drug: Sorafenib; Drug: Myeloid Growth Factor; Procedure: Lymph Node Sampling; Drug: ^1^1C-methionine
- High-Risk (Experimental): Lymph node sampling takes place pretreatment and pre-surgery. Participants receive 6 weeks (2 cycles) chemotherapy (vincristine and irinotecan). The tumor is evaluated for treatment response. 3 cycles of chemotherapy [vincristine, doxorubicin, cyclophosphamide/ifosfamide, etoposide (or etoposide phosphate) (VDC/IE)] are given. Dexrazoxane is given prior to each dose of doxorubicin. Radiation therapy begins at week 4 or 20 (depending on tumor location) while receiving vincristine and irinotecan. 2 cycles of VDC/IE, 4 cycles of modified vincristine, dactinomycin, cyclophosphamide (VAC), then 2 cycles of modified vincristine/irinotecan (total of 54 weeks). High risk participants also receive additional maintenance therapy beginning week 55 with anti-angiogenic chemotherapy (bevacizumab, sorafenib, cyclophosphamide). Myeloid growth factor is given as needed.
  Participants also receive ^1^1C-methionine as described in the intervention section.
  Interventions: Drug: Vincristine; Drug: Dactinomycin; Drug: Cyclophosphamide; Procedure: Surgical Resection; Procedure: Radiation; Drug: Bevacizumab; Drug: Sorafenib; Drug: Myeloid Growth Factor; Procedure: Lymph Node Sampling; Drug: Irinotecan; Drug: Ifosfamide; Drug: Etoposide; Drug: Etoposide Phosphate; Drug: Doxorubicin; Drug: Dexrazoxane; Drug: ^1^1C-methionine

INTERVENTIONS:
Drug: Vincristine — Dosage and route of administration:
  * < 1 year of age=0.025 mg/kg intravenously (IV)
  * > 1 year and < 3 years= 0.05 mg/kg IV
  * ≥ 3 years=1.5 mg/m^2 IV. Maximum dose 2 mg in all participants.
  Other Names: Oncovin®
Drug: Dactinomycin — Dosage and route of administration:
  * < 1 year=0.025 mg/kg IV push
  * ≥ 1 year=0.045 mg/kg IV push over 1 to 5 minutes.
  Other Names: Actinomycin-D; Cosmegen®
Drug: Cyclophosphamide — Dosage and route of administration:
  During VAC chemotherapy:
  * < 3 years of age = 40 mg/kg IV
  * ≥ 3 years of age = 1200 mg/m^2 IV, with MESNA.
  During maintenance for intermediate-risk participants:
  * oral cyclophosphamide 50 mg/m^2/dose/day (liquid or tablet)
  Other Names: Cytoxan(R)
Procedure: Surgical Resection — Surgery will be performed for the primary site tumor with the goal of removing tumor cells while maintaining function in the organ or adjacent organs involved.
  Other Names: Surgery
  Arms: High-Risk; Intermediate-Risk; Low-Risk, Subset 1
Procedure: Radiation — Radiation therapy will be delivered at approximately week 13 (intermediate risk) or week 19 (high risk) after initiation of chemotherapy. Certain patients will receive radiation at week 4.
  Other Names: Proton Beam Radiation; External Beam Radiation; Brachytherapy
Drug: Bevacizumab — Dosage and route of administration: 15 mg/kg/dose/day IV.
  Other Names: rhuMab; VEGF; Avastin®
  Arms: High-Risk; Intermediate-Risk
Drug: Sorafenib — Dosage and route of administration: 90 mg/m^2/dose twice daily.
  Other Names: Nexavar®
  Arms: High-Risk; Intermediate-Risk
Drug: Myeloid Growth Factor — If a participant's chemotherapy has been delayed or modified for hematologic toxicity, or if participant experiences a significant life-threatening toxicity due to bone marrow suppression, myeloid growth factor (either filgrastim or peg-filgrastim) will be given per institutional practice.
  High Risk participants receive filgrastim 5 micrograms/kg/day (maximum 300 micrograms) subcutaneously beginning 24-36 hours after the last dose of chemotherapy. Continue at least 7 days, or until the ANC ≥750/µL whichever comes last. Sargramostim or peg-filgrastim may not be used.
  Other Names: G-CSF; Filgrastim; Pegfilgrastim
Procedure: Lymph Node Sampling — Clinical and/or imaging evaluation of regional lymph nodes will be conducted pretreatment and preoperatively as part of staging. This will aid in determining the efficacy of this procedure in defining involved lymphatics in "at risk" patients.
Drug: Irinotecan — Dosage and Route Administration: During interval compressed therapy - irinotecan 50mg/m^2 IV (maximum dose 100 mg/day) daily x 5.
  Other Names: Camptosar ®
  Arms: High-Risk
Drug: Ifosfamide — Dosage and Route of Administration: During interval compressed therapy - Age > 1 year: 1800 mg/m^2/day IV x 5 Age <1 year: treat with 50% doses calculated on a m^2 basis.
  Other Names: Ifex ®
  Arms: High-Risk
Drug: Etoposide — Dosage and Route of Administration:
  Age >1 year 100 mg/m^2/day IV x 5 Age < 1 year treat with 50% doses calculated on a m^2 basis
  Other Names: VP-16; Vepesid®
  Arms: High-Risk
Drug: Etoposide Phosphate — Dosage and Route of Administration: Used in substitution for etoposide in participants who experience allergic reaction. It will be administered 100 mg/m^2/day IV.
  Other Names: Etopophos®
  Arms: High-Risk
Drug: Doxorubicin — Dosage and route of Administration:
  Age ≥1 year, 37.5 mg/m^2 IV over 1 hour x 2 days Age <1 year, 18.75 mg/m^2 (i.e., a 50% dose reduction) IV over 1 hour x 2 days.
  Other Names: Adriamycin®
  Arms: High-Risk
Drug: Dexrazoxane — Dosage and Route of Administration: Dexrazoxane dose should be 10x that of doxorubicin.
  Age ≥1 year, 375 mg/m^2 IV over 15-30 minutes Age <1 year, 187l.5 mg/m^2 (i.e., a 50% dose reduction) IV over 15-30 minutes.
  Other Names: Zinecard
  Arms: High-Risk
Drug: ^1^1C-methionine — Participants receive ^1^1C-methionine to relate the distribution, intensity and change in ^1^1C-methionine CTPET imaging of the primary site to tumor control and patient outcome.
  Other Names: Contrast Media

SUMMARY:
This study will treat participants with newly diagnosed, low, intermediate and high risk rhabdomyosarcoma (RMS) using multi-modality risk-adapted therapy with standard or intensified dose chemotherapy, radiation and surgical resection. Intermediate and high risk participants will receive an additional 12 weeks (4 cycles) of maintenance therapy with anti-angiogenic chemotherapy.

PRIMARY OBJECTIVE:

* Estimate event-free survival for intermediate risk participants treated with vincristine, dactinomycin and cyclophosphamide with the addition of maintenance anti-angiogenic therapy.

SECONDARY OBJECTIVES:

* Estimate the false negative rate and incidence of additional positive lymph nodes in participants undergoing sentinel lymph node biopsy followed by limited nodal dissection.
* Maintain a high local control rate in participants treated with surgery and/or limited volume proton and photon radiation without dose escalation.
* Define the incidence and type of failure in participants who receive risk-adapted local therapy relative to the primary tumor volume.
* Establish the feasibility of delivering 4 cycles of maintenance anti-angiogenic chemotherapy in intermediate and high risk patients following standard chemotherapy.
* Estimate the event free survival for high risk patients receiving interval dose compressed therapy and maintenance anti-angiogenic therapy.
* Define the incidence of CTC grade 3 and higher toxicities (and specific grade 1-2 toxicities) related to proton beam therapy.

DETAILED DESCRIPTION:
Participants will be stratified based on both a pretreatment staging system and a post-surgery surgico/pathologic clinical grouping system. Treatment for low-risk (subset 1) participants will consist of chemotherapy and radiation. Low-risk (subset 2) and intermediate-risk participants will receive chemotherapy and radiation and/or undergo surgery to destroy/remove the tumor. Intermediate-risk participants will also receive 16 weeks of maintenance chemotherapy. High-risk participants will receive chemotherapy and radiation therapy. High-risk participants will also receive additional maintenance therapy with anti-angiogenic chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed participants with localized rhabdomyosarcoma (RMS).
* Must have either low-, intermediate-, or high-risk disease, defined as:

  * Low-risk: Embryonal, botryoid, spindle cell tumors only (Subset 1: Stage 1, Group I; Stage 1 Group I; Stage 1 Group III orbital only; Stage 2 Group I; Stage 2 Group II) (Subset 2: Stage 1 Group III non orbit; Stage 3 Group I, II)
  * Intermediate-risk: Embryonal, botryoid, or spindle cell RMS Stage 2 or 3 and Group III; Alveolar, undifferentiated, or anaplastic RMS: Stage 1-3, group I-I; I)
  * High-risk: Embryonal, botryoid, spindle cell, alveolar, undifferentiated, or anaplastic RMS with metastatic disease at diagnosis (stage 4).
  * Participants treated on this protocol in the low or intermediate risk arm who experience disease progression prior to week 13 will transfer to the high risk arm and proceed with high risk chemotherapy starting at week 1 of the protocol.
* Age < 22 years (eligible until 22nd birthday)
* Performance level corresponding to ECOG score of 0, 1, or 2. The Lansky performance score should be used for participants < 16 years
* Participant has received no prior radiotherapy or chemotherapy for rhabdomyosarcoma (excluding steroids) unless an emergency situation requires local tumor treatment. Prior biopsy, surgical resection and lymph node sampling is allowed.
* Initiation of chemotherapy is planned within 6 weeks (42 days) of the definitive biopsy or surgical resection.
* Adequate bone marrow function defined as:

  * Peripheral absolute neutrophil count (ANC) ≥ 750/μL
  * Platelet count ≥ 75,000/μL (transfusion independent)
* Adequate liver function defined as total bilirubin ≤ 1.5 x upper limit of normal (ULN) for age. Participants with biliary or hepatic primaries with bilirubin values greater than 1.5 x ULN may be enrolled on study if all other eligibility criteria are met.
* Adequate renal function defined as:

  * Creatinine clearance or radioisotope GFR ≥ 70 mL/min/1.732 or
  * Serum creatinine based on age and gender
  * Participants with urinary tract obstruction by tumor must meet the renal function criteria listed above AND must have unimpeded urinary flow established via decompression of the obstructed portion of the urinary tract.
* Patients requiring emergency radiation therapy are eligible for enrollment on this study.
* Females of child-bearing potential cannot be pregnant or breast-feeding. Female participants ≥ 10 years of age or post-menarchal must have a negative serum or urine pregnancy test within 24 hours prior to beginning treatment. Female participants who are breast feeding must agree to stop breast feeding.
* Sexually active patients of childbearing potential must be willing to use effective contraception during therapy and for at least 1 month after treatment is completed.
* No evidence of active, uncontrolled infection.
* All participants and/or their parents or legal guardians must sign a written informed consent.

Exclusion Criteria:

* Participants who fail to meet one or more of the inclusion criteria will be excluded.

Inclusion Criteria for Contrast-Enhanced Ultrasound (CEUS) Sub-Study:

* Newly diagnosis or suspected diagnosis of previously untreated participants with rhabdomyosarcoma (RMS). NOTE: Patients with suspected diagnosis of RMS may enroll on screening part of study but must have histologic diagnosis to enroll on treatment part of study.
* Must have either intermediate-risk or high risk disease.
* 0-21 years of age.

Exclusion Criterial for CEUS Sub-Study:

* Undergoing upfront surgical resection of the primary tumor.
* History of allergy to Optison(TM) contrast agent or blood products.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 115 (Actual)
Dates: Start 2013-12-04 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2030-06 (Estimated)

PRIMARY OUTCOMES:
Event-free survival (intermediate risk arm) | 2 years after last intermediate risk arm enrollment
  To estimate event-free survival for intermediate risk participants treated by vincristine-dactinomycin-cyclophosphamide (VAC) with the addition of maintenance anti-angiogenic therapy

SECONDARY OUTCOMES:
Event-free survival (high risk arm) | 5 years after last high-risk arm enrollment
  To estimate event-free survival for high risk participants.
Rate of false negative and false positive the sentinel lymph node procedure (low and intermediate risk arms) | 2 years after last low or intermediate arm enrollment
  Estimate the false negative rate and incidence of additional positive lymph nodes in participants undergoing sentinel lymph node biopsy followed by limited nodal dissection.
Rate of false negative and false positive the sentinel lymph node procedure (high risk arm) | 5 years after last high risk arm enrollment
  Estimate the false negative rate and incidence of additional positive lymph nodes in participants undergoing sentinel lymph node biopsy followed by limited nodal dissection.
Local failure rate (low and intermediate risk arms) | 2 years after last low or intermediate risk arm enrollment
  Maintain a high local control rate in participants treated with surgery and / or limited volume proton and photon radiation without dose escalation
Local failure rate (high risk arm) | 5 years after last high risk arm enrollment
  Maintain a high local control rate in participants treated with surgery and / or limited volume proton and photon radiation without dose escalation
Patterns of failure (low and intermediate risk arms) | 2 years after last low or intermediate risk arm enrollment
  Define the incidence and type of failure in participants who receive risk-adapted local therapy relative to the primary tumor volume
Patterns of failure (high risk arm) | 5 years after last high risk arm enrollment
  Define the incidence and type of failure in participants who receive risk-adapted local therapy relative to the primary tumor volume
Number of patients that complete all cycles of maintenance chemotherapy (intermediate risk arm) | 2 years after last low or intermediate risk arm enrollment
  Establish the feasibility of delivering 4 cycles of maintenance antiangiogenic chemotherapy (bevacizumab / sorafenib / low dose cyclophosphamide) in intermediate risk patients following standard chemotherapy.
Number of patients that complete all cycles of maintenance chemotherapy (high risk arm) | 5 years after last high risk arm enrollment
  Establish the feasibility of delivering 4 cycles of maintenance antiangiogenic chemotherapy (bevacizumab / sorafenib / low dose cyclophosphamide) in high risk patients following standard chemotherapy.
Incidence of CTC grade 3 and higher toxicities related to proton bream therapy (low and intermediate and high risk arms) | 2 years after last enrollment
  Define the incidence of CTC grade 3 and higher toxicities (and specific grade 1-2 toxicities) related to proton beam therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew J. Krasin, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (4):
- United States (4):
  - University of Florida Proton Therapy Institute, Jacksonville, Florida
  - Nemours Children's Clinic, Jacksonville, Florida
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Cook Children's Medical Center, Fort Worth, Texas

REFERENCES:
- [Derived] Patel AG, Chen X, Huang X, Clay MR, Komorova N, Krasin MJ, Pappo A, Tillman H, Orr BA, McEvoy J, Gordon B, Blankenship K, Reilly C, Zhou X, Norrie JL, Karlstrom A, Yu J, Wodarz D, Stewart E, Dyer MA. The myogenesis program drives clonal selection and drug resistance in rhabdomyosarcoma. Dev Cell. 2022 May 23;57(10):1226-1240.e8. doi: 10.1016/j.devcel.2022.04.003. Epub 2022 Apr 27. PMID 35483358
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols